CLINICAL TRIAL: NCT00144820
Title: Intra-Articular Injections of Hyaluronan Versus 20 Ml NaCl Versus Placebo in Treatment of Knee Osteoarthritis: a Randomised, Double-Blind, Placebo Controlled Single Centre Trial.
Brief Title: Hyaluronan Versus NaCl 20 Ml Versus Placebo in Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA 99005gs
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Hyaluronan; Gonarthrosis; Osteoarthritis,knee; Double-blinded; Placebo controlled; Randomised
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

INTERVENTIONS:
Drug: Injection of Hyaluronan or Saline

SUMMARY:
251 consecutive patients with knee arthrosis were randomized to one of three interventions: Four weekly injections of 2 ml isotonic saline (placebo), 2 ml sodium hyaluronate (hyaluronan) or 20 ml isotonic saline (excessive saline).

They all suffered from clinically and radiologically verified arthrosis of the knee with daily pain that did not respond to treatment with analgetics.

Results were evaluated at weeks 1,2,3,4,8,12,16 and 26. Biochemical markers for bone and cartilage degradation were measured in urine/blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients, men/women age > 60 years with clinical,
* Radiological and possible arthroscopical verified knee osteoarthritis.
* Knee pain on the day of examination scoring more than 20 mm on a visual analogue scale (VAS) at baseline.

Exclusion Criteria:

* Age below 60
* Unconsciousness
* Psychosis
* Demens
* Ingestion of drugs that may influence the results of the clinical examinations
* Inflammatory diseases of the joints
* Rheumatoid arthritis or other inflammatory arthritis as diagnosed by American College of Rheumatology criteria
* Contraindication to hyalgan treatment
* Previous intraarticular fracture of a knee joint
* Infection or skin disease located at the place of injection and invasive procedures done to the knee joint within previous two months inclusive intra-articular injections of steroids.
* Any other condition that might interfere with the efficacy assessment or completion of the trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251
Dates: Start 1999-05; Study Completion 2001-11

PRIMARY OUTCOMES:
Pain measured on a visual scale on movement (VAS-movement)
At rest (VAS-rest)
During the night (VAS-night)

SECONDARY OUTCOMES:
KOOS scores (knee injury and osteoarthritis outcome score)
Daily consumption of analgetics
Cartilage and bone degradation markers
The quadriceps circumference (cm), ability to bend (degrees flexion) and stretch (degrees extension) the knee joint
Global assessment patient
Global assessment investigator

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lundsgaard, MD, Principal Investigator — Copenhagen Trial Unit (CTU)
Locations (1):
- Copenhagen Trial Unit, H:S Rigshospitalet. dept. 7102, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Lundsgaard C, Dufour N, Fallentin E, Winkel P, Gluud C. Intra-articular sodium hyaluronate 2 mL versus physiological saline 20 mL versus physiological saline 2 mL for painful knee osteoarthritis: a randomized clinical trial. Scand J Rheumatol. 2008 Mar-Apr;37(2):142-50. doi: 10.1080/03009740701813103. PMID 18415773